CLINICAL TRIAL: NCT04692025
Title: A Randomized, Single Center, Open-label, Phase I Study to Evaluate the Effect of Food and Fasting on the Pharmacokinetics of ASC41 Tablets in Healthy Volunteers
Brief Title: Study to Evaluate the Effect of Food on the Pharmacokinetics of ASC41 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gannex Pharma Co., Ltd. (Industry)
Collaborators: Hunan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASC41-103
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy; NAFLD; Hyperlipidemia
Keywords: Healthy Volunteers; NAFLD; NASH; Hyperlipidemia; LDL-C
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): ASC41 one tablet, on Day 1 before meal；ASC41 one tablet, on Day 15 after meal.
  Interventions: Drug: ASC41 tablet
- Group 2 (Experimental): ASC41 one tablet, on Day 1 after meal；ASC41 one tablet, on Day 15 before meal.
  Interventions: Drug: ASC41 tablet

INTERVENTIONS:
Drug: ASC41 tablet — Oral tablet

SUMMARY:
This study is to evaluate the effect of food on the pharmacokinetics of a single dose of ASC41 tablet in healthy volunteers, comparing fasting and postprandial pharmacokinetic parameters of Tmax, Cmax, AUC0-t, AUC0-∞.

ELIGIBILITY:
Key Inclusion Criteria:

* 19kg/m2 ≤ BMI <40kg/m2.

Key Exclusion Criteria:

* A history of thyroid disease.
* History of, or current liver disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-27 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
AUC of ASC41 | Up to 19 days
  Evaluate the Area under the plasma concentration versus time curve after single oral dose of ASC41 administered to healthy volunteers.
Cmax of ASC41 | Up to 19 days
  Evaluate the Peak Plasma Concentration after single oral dose of ASC41 administered to healthy volunteers.

SECONDARY OUTCOMES:
t1/2 of ASC41 | Up to 19 days
  Evaluate the Terminal-Phase Half-Life after single oral dose of ASC41 administered to healthy volunteers.
CL/F of ASC41 | Up to 19 days
  Evaluate the Apparent Systemic Clearance after single oral dose of ASC41 administered to healthy volunteers.
Vd/F of ASC41 | Up to 19 days
  Evaluate the Apparent Volume of Distribution after single oral dose of ASC41 administered to healthy volunteers.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 19 days
  Occurrence of Serious Adverse Event (SAE), Adverse Event (AE) resulting in treatment discontinuation and/or dose reductions, and AE of special interest, from baseline up to 19 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan provincial people's hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided